CLINICAL TRIAL: NCT02128685
Title: A Randomized Double-blind Controlled Trial of Use of Dydrogesterone in Women With Threatened Miscarriage in the First Trimester
Brief Title: Randomized Double-blind Controlled Trial of Use of Dydrogesterone in Threatened Miscarriage
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Diana Man-Ka Chan, Resident, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UW 13-292
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-10

CONDITIONS: Pregnancy
Keywords: Threatened miscarriage; Dydrogesterone; Randomized controlled trial
MeSH Terms: conditions — Abortion, Threatened | interventions — Dydrogesterone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Dydrogesterone (Active Comparator): Patients allocated to the dydrogesterone group will receive oral dydrogesterone 40mg stat, followed by 10mg orally three times a day, and placebo will be used in the control group accordingly. Patients will be followed up with weekly pelvic ultrasound till 12 completed weeks of gestation or 1 week after the bleeding stopped, whichever is longer.
  Interventions: Drug: Dydrogesterone
- Placebo pill (Placebo Comparator): Patients allocated to the dydrogesterone group will receive oral dydrogesterone 40mg stat, followed by 10mg orally three times a day, and placebo will be used in the control group accordingly. Patients will be followed up with weekly pelvic ultrasound till 12 completed weeks of gestation or 1 week after the bleeding stopped, whichever is longer.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dydrogesterone
  Other Names: Duphaston
  Arms: Dydrogesterone
Drug: Placebo
  Arms: Placebo pill

SUMMARY:
The aim of this study is to determine whether the dydrogesterone therapy is associated with reduction in miscarriage in women with first trimester threatened miscarriage. The hypothesis is that the dydrogesterone therapy will significantly reduce the risk of miscarriage in women with threatened miscarriage.

ELIGIBILITY:
Inclusion Criteria:

* Age of women from 18-40 years at the time of recruitment (not beyond 40th birthday)
* Absence of fever
* Gestation less than 12 completed weeks as defined by pelvic ultrasound
* Presence of intrauterine gestational sac(s) if an urine pregnancy test is first positive within past 2 weeks
* Presence of intrauterine fetus(es) with crown-rump length of <7mm and no fetal pulsation, or presence of intrauterine fetus(es) with positive fetal heart pulsation confirmed on pelvic scanning

Exclusion Criteria:

* Age of women >40 years at the time of recruitment
* History of recurrent miscarriage defined as at least three consecutive spontaneous miscarriages
* History of known parental chromosomal abnormalities
* Heavy vaginal bleeding requiring surgical intervention
* Severe abdominal pain requiring surgical intervention
* Absence of cardiac pulsation in a fetal pole with crown-rump length of >=7mm on transvaginal scanning
* Use of hCG or progesterone treatment for threatened miscarriage prior to recruitment

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 406 (Actual)
Dates: Start 2016-03; Primary Completion 2018-05-31 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
The chance of miscarriage before 20 weeks of gestation | At 20 weeks of gestation

SECONDARY OUTCOMES:
Live birth rate | At the time of delivery, from 24 weeks of gestation till term gestation
The proportion of heavy vaginal bleeding or severe abdominal pain requiring surgical intervention (<20 weeks) | Before 20 weeks of gestation
The incidence of antepartum hemorrhage | From 24 weeks of gestation till term
  Any vaginal bleeding during pregnancy from the 24th week gestational age to term
The incidence of placenta previa | From 24 weeks of gestation till term
  Placenta is being inserted partially or wholly in the lower uterine segment and will be diagnosed by antenatal ultrasound at second and third trimesters
The incidence of pregnancy-induced hypertension | From 20 weeks of gestation till term
  Any development of newly-onset hypertension (blood pressure persistently >=140/90mmHg on two occasions at least 4 hours apart) during pregnancy after 20 weeks gestation, labour or the puerperium in a previously normotensive non-proteinuric women
The incidence of intrauterine death | After 24 weeks of gestation till term
  Fetus dies in uterus after 24 weeks gestation
The incidence of preterm labour | From 24 weeks to 36 weeks gestation
  Any premature spontaneous delivery from 24 weeks to 36 weeks gestation
Low birth weight at term (grams) | After 37 weeks gestation
  Baby born with birth weight less than 2500g at or after 37 weeks gestation

CONTACTS AND LOCATIONS:
Overall Officials: Man Ka Diana Chan, MBBS(HK), Principal Investigator — Department of Obstetrics & Gynaecology, Queen Mary Hospital
Locations (3):
- Hong Kong (3):
  - Department of Obstetrics and Gynaecology, PYNEH, Chai Wan
  - Department of Obstetrics & Gynaecology, Queen Mary Hospital, Hong Kong
  - Department of Obstetrics & Gynaecology, Kwong Wah Hospital, Mong Kok

REFERENCES:
- [Derived] Chan DMK, Cheung KW, Ko JKY, Yung SSF, Lai SF, Lam MT, Ng DYT, Lee VCY, Li RHW, Ng EHY. Use of oral progestogen in women with threatened miscarriage in the first trimester: a randomized double-blind controlled trial. Hum Reprod. 2021 Feb 18;36(3):587-595. doi: 10.1093/humrep/deaa327. PMID 33331637
- [Derived] Chan DM, Cheung KW, Yung SS, Lee VC, Li RH, Ng EH. A randomized double-blind controlled trial of the use of dydrogesterone in women with threatened miscarriage in the first trimester: study protocol for a randomized controlled trial. Trials. 2016 Aug 17;17(1):408. doi: 10.1186/s13063-016-1509-8. PMID 27534747